CLINICAL TRIAL: NCT05926180
Title: A Phase 1, Open-label, Non-Randomized Study to Assess the Effect of DZD9008 on the Pharmacokinetics of the Cocktail Probes Representative for CYP3A4, P-gp, BCRP and OATP1B1 in Patients with EGFR or HER2 Mutant Advanced Non-small Cell Lung Cancer
Brief Title: Assessing the Effect of DZD9008 on the Pharmacokinetics of the Cocktail Probes Representative for CYP3A4, P-gp, BCRP and OATP1B1 in Patients with EGFR or HER2 Mutant Advanced Non-small Cell Lung Cancer (WU-KONG19)
Status: Completed | Phase: Phase 1 | Type: Interventional
Sponsor: Dizal Pharmaceuticals (Industry)
Responsible Party: Sponsor
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Treatment
Other Study IDs: DZ2021E0009
Record Dates: First submitted 2023-06-22; First posted 2023-07-03 (Actual); Last update posted 2024-12-13 (Actual); Status verified 2024-12

CONDITIONS: Non-small Cell Lung Cancer
MeSH Terms: conditions — Carcinoma, Non-Small-Cell Lung | interventions — Midazolam; Digoxin; Rosuvastatin Calcium

STUDY DESIGN:
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: Yes | FDA-regulated Device: No | US Export: No

ARMS (1):
- DZD9008 + Probe Drugs (Experimental): Single dose of 2 mg midazolam (oral solution), 0.25 mg digoxin (tablet) and 10mg rosuvastatin (tablet) and in combination with 300 mg DZD9008 (tablet)
  Interventions: Drug: DZD9008 and Probe drugs (midazolam, digoxin, rosuvastatin)

INTERVENTIONS:
Drug: DZD9008 and Probe drugs (midazolam, digoxin, rosuvastatin) — Patients will receive single oral doses of probe drugs alone and after at least 27 days of treatment with DZD9008, 300 mg, once daily, until a treatment discontinuation criterion is met. Each patient will receive a single oral dose of DZD9008 on Day 7, and DZD9008 once daily for 27 days from Day 9 to Day 35. Patients will also receive a single oral dose of 2 mg midazolam on Day 1 and Day 32, and oral dose of 10 mg rosuvastatin and 0.25 mg digoxin cocktail on Day 2, Day 7 and Day 33.
  Other Names: Inapplicable

SUMMARY:
This study will treat patients with advanced NSCLC who have progressed following prior therapy in order to assess the effect of DZD9008 on exposure of midazolam, digoxin and rosuvastatin, through multiple PK parameters, when administrated as a single dose alone and in combination with DZD9008. Also, it will assess the safety and tolerability of DZD9008 in the presence and absence of co-administration of cocktail probes.

ELIGIBILITY:
Inclusion Criteria:

* Aged at least 18 years old, be able to provide a signed and dated, written informed consent.
* Patients must have documented histologically or cytologically confirmed locally advanced or metastatic NSCLC with EGFR or HER2 mutations and have progressed from, been refractory to or are intolerant to prior standard therapy without preferred alternative therapy.
* Eastern Cooperative Oncology Group (ECOG) performance status 0 - 1 at ICF signature with no deterioration over the previous 2 weeks.
* Predicted life expectancy ≥ 12 weeks

Exclusion Criteria:

* Patients with a known hypersensitivity to DZD9008, rosuvastatin, digoxin, midazolam, or any of the excipients of the products.
* Concomitant medication or any clinical condition contraindicated for use with rosuvastatin, digoxin, midazolam.
* Major surgery (excluding placement of vascular access) within 4 weeks of the first dose of study treatment.
* Patients currently receiving (or unable to stop use prior to receiving the first dose of study treatment) medications or herbal supplements known to be potent inhibitors or inducers of CYP3A4, BCRP, OATP1B1 and P-gp.
* Patients who have BCRP (ABCG2) polymorphism c.421C>A (p.Q141K, rs2231142).
* Patients with previous allogenic bone marrow transplant or non-leukocyte depleted whole blood transfusion within 120 days of the date of the genetic sample collection.
* Patients with liver metastases, spinal cord compression or leptomeningeal metastasis.
* Any evidence of severe or uncontrolled systemic diseases, including uncontrolled hypertension and active bleeding diatheses.
* Participants with active infection including but not limited to hepatitis B virus (HBV), hepatitis C virus (HCV), human immunodeficiency virus (HIV) (refer to CSP) and active infection of COVID-19.
* Inadequate bone marrow reserve or organ function.
* Past medical history of interstitial lung disease, drug-induced interstitial lung disease, radiation pneumonitis which required steroid treatment, or any evidence of clinically active interstitial lung disease.
* Refractory nausea and vomiting, chronic gastrointestinal diseases, inability to swallow the formulated product or previous significant bowel resection that would preclude adequate absorption of study treatment.
* Women who are pregnant or breast feeding.
* Known history of bleeding diathesis, i.e., hemophilia, Von Willebrand disease.
* History of stroke or intracranial haemorrhage within 6 months

Other protocol-defined inclusion/exclusion criteria may apply.

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 25 (Actual)
Dates: Start 2023-07-31 (Actual); Primary Completion 2024-05-16 (Actual); Study Completion 2024-09-28 (Actual)

PRIMARY OUTCOMES:
Cmax of midazolam, 1-OH Midazolam, digoxin and rosuvastatin alone and in combination with DZD9008 | Days 1-35
AUC0-t of midazolam, 1-OH Midazolam, digoxin and rosuvastatin alone and in combination with DZD9008 | Days 1-35
Ratio of AUC of midazolam, 1-OH midazolam, digoxin and rosuvastatin between substrate alone and with DZD9008 | Days 1-35
Ratio of Cmax of midazolam, 1-OH midazolam, digoxin and rosuvastatin between substrate alone and with DZD9008 | Days 1-35
AUC0-inf of midazolam, 1-OH Midazolam, digoxin and rosuvastatin alone and in combination with DZD9008, if applicable | Days 1-35

CONTACTS AND LOCATIONS:
Locations (1):
- Shandong Cancer Hospital (Shandong Provincial Institute of Cancer Prevention and Treatment), Jinan, Shandong, China

IPD SHARING:
Plan to Share IPD: No